CLINICAL TRIAL: NCT00111540
Title: An Open Label Study to Examine the Long Term Effect on Glucose Control (HbA1c) and Safety and Tolerability of Exenatide Given Two Times a Day to Subjects With Type 2 Diabetes Mellitus
Brief Title: Study to Examine the Effect on Glucose Control and Safety/Tolerability of Exenatide Given Two Times a Day to Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2993-119
Record Dates: First submitted 2005-05-23; First posted 2005-05-24 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: exenatide; diabetes; Amylin; exendin-4
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exenatide (Experimental): Exenatide 5 mcg for 4 weeks (transition) then 10 mcg to study termination
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5 mcg, twice a day for 4 weeks (transition period), then 10 mcg twice a day till study termination
  Other Names: Byetta; exendin-4; AC2993

SUMMARY:
This open label study is designed to assess long term glucose control, as measured by hemoglobin A1c (HbA1c) and to evaluate long term safety and tolerability in subjects with type 2 diabetes mellitus who receive subcutaneously injected exenatide administered twice a day.

ELIGIBILITY:
Inclusion Criteria:

* The subject has an HbA1c value <=11.0%
* The subject has a body mass index (BMI) of 25 kg/m^2 to 45 kg/m^2, inclusive

Exclusion Criteria:

* Is currently treated with certain medications, including exogenous insulin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2002-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Visit 1 to each protocol visit | Day 1, Weeks 2, 4, 8, 15, 22, 30, 38, 46 and every 12 weeks while on study (78 week target)
  Change in HbA1c from Visit 1 to each visit up to open-ended study termination
Change in body weight from Visit 1 to each protocol visit | Day 1, Weeks 2, 4, 8, 15, 22, 30, 38, 46 and every 12 weeks while on study (78 week target)
  Change in body weight (kg) from Visit 1 to each visit up to open-ended study termination
Change in fasting plasma glucose from Visit 1 to each protocol visit | Day 1, Weeks 2, 4, 8, 15, 22, 30, 38, 46 and every 12 weeks while on study (78 week target)
  Change in fasting plasma glucose from Visit 1 to each visit up to open-ended study termination
Change in lipids from Visit 1 to each protocol visit | Day 1, Weeks 2, 4, 8, 15, 22, 30, 38, 46 and every 12 weeks while on study (78 week target)
  Change in lipids from Visit 1 to each visit up to open-ended study termination

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (60):
- United States (60):
  - Research Site, Birmingham, Alabama
  - Research Site, Anaheim, California
  - Research Site, Bellflower, California
  - Research Site, Burlingame, California
  - Research Site, Chula Vista, California
  - Research Site, Concord, California
  - Research Site, Encino, California
  - Research Site, Fremont, California
  - Research Site, La Jolla, California
  - Research Site, Los Gatos, California
  - Research Site, Moreno Valley, California
  - Research Site, Redwood City, California
  - Research Site, San Mateo, California
  - Research Site, Walnut Creek, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Largo, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Blairsville, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Gulfport, Mississippi
  - Research Site, Picayune, Mississippi
  - Research Site, Chesterfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Cary, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Mentor, Ohio
  - Research Site, Clinton, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Midland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Olympia, Washington
  - Research Site, Spokane, Washington

REFERENCES:
- [Result] Blonde L, Klein EJ, Han J, Zhang B, Mac SM, Poon TH, Taylor KL, Trautmann ME, Kim DD, Kendall DM. Interim analysis of the effects of exenatide treatment on A1C, weight and cardiovascular risk factors over 82 weeks in 314 overweight patients with type 2 diabetes. Diabetes Obes Metab. 2006 Jul;8(4):436-47. doi: 10.1111/j.1463-1326.2006.00602.x. PMID 16776751
- [Result] Buse JB, Klonoff DC, Nielsen LL, Guan X, Bowlus CL, Holcombe JH, Maggs DG, Wintle ME. Metabolic effects of two years of exenatide treatment on diabetes, obesity, and hepatic biomarkers in patients with type 2 diabetes: an interim analysis of data from the open-label, uncontrolled extension of three double-blind, placebo-controlled trials. Clin Ther. 2007 Jan;29(1):139-53. doi: 10.1016/j.clinthera.2007.01.015. PMID 17379054
- [Result] Klonoff DC, Buse JB, Nielsen LL, Guan X, Bowlus CL, Holcombe JH, Wintle ME, Maggs DG. Exenatide effects on diabetes, obesity, cardiovascular risk factors and hepatic biomarkers in patients with type 2 diabetes treated for at least 3 years. Curr Med Res Opin. 2008 Jan;24(1):275-86. doi: 10.1185/030079908x253870. PMID 18053320
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Derived] Nelson P, Poon T, Guan X, Schnabel C, Wintle M, Fineman M. The incretin mimetic exenatide as a monotherapy in patients with type 2 diabetes. Diabetes Technol Ther. 2007 Aug;9(4):317-26. doi: 10.1089/dia.2006.0024. PMID 17705687